CLINICAL TRIAL: NCT01911858
Title: Non-controlled Prospective Cohort Study of the Use of Askina® Calgitrol® Paste on III Degree Burns in Adults
Brief Title: Askina Calgitrol Paste Burns
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: BBraun Medical SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: OPM-G-H-1204
Record Dates: First submitted 2013-07-25; First posted 2013-07-30 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Third Degree Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Askina Calgitrol Paste (Experimental)
  Interventions: Device: Askina Calgitrol Paste

INTERVENTIONS:
Device: Askina Calgitrol Paste

SUMMARY:
The purpose of the study is to demonstrate that Askina® Calgitrol® Paste is safe to use on III degree burns by quantifying the concentration of silver in the blood during treatment and thus to show that the amount of silver absorbed will be no greater than those reported in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥>18 years age). No upper age limit
* III degree thermal burns from 2-30% TBSA as determined by the Rule of Nines
* Patients who underwent initial treatment within 24 hours after the injury at the latest
* Patients who underwent initial treatment directly at the Burn Centre of FNKV or the initial treatment was in accordance with the standard of care of the Centre
* All patients will have been hospitalised
* Patients who are capable of giving signing informed consent and have done so.

Exclusion Criteria:

* Patients with electrical or chemical burns
* Patients with already infected wounds
* Patients taking systemic antibiotics on admission
* Patients pregnant or lactating
* Patients who fall into "vulnerable population" group with respect to informed consent or who are not capable of giving informed consent
* Patients who used or were treated with silver products for other reasons than treatment of the acute burn in the last 3 months
* Patients whose other burn wounds are being treated with silver products.
* Patients receiving renal dialysis
* Known allergy or sensitivity to any of the ingredients in Askina® Calgitrol® Paste.
* Simultaneous participation in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The quantification of the amount of silver found in plasma during the treatment | Change from Baseline in Blood at 3 days
The quantification of the amount of silver found in plasma during the treatment | Change from Baseline in Blood immediately after the removal of the last investigational dressing (the day before necrotomy, an expected average between 3-10 days after inclusion)

SECONDARY OUTCOMES:
Wound bed and periwound skin conditions | At each dressing change (an expected average of one day)
  Data will not be recorded at specific time points due to individual changing patterns. The investigator will make a subjective description of the wound bed covered by necrosis, slough/fibrin, granulation tissue and epithelialisation and by the condition of the peri-wound skin.
Clinical signs of infection | At each dressing change (an expected average of one day)
  Data will not be recorded at specific time points due to individual changing patterns.
  The presence and intensity of clinical signs of infection will be assessed at the start of the study and at each dressing change using clinical judgment and a scoring system modified from the one published by Trial and al.
Patient comfort | At each dressing change (an expected average of one day)
  Data will not be recorded at specific time points due to individual changing patterns.
  The investigator will complete a Likert scale score (1-4, Poor, Fair, Good, Excellent) for each ease of application and ease of removal of Askina Calgitrol Paste at each dressing change.
Number of dressing changes | At each dressing change (an expected average of one day)
  Data will not be recorded at specific time points due to individual changing patterns.
Adverse Events or Adverse device related event | At each dressing change